CLINICAL TRIAL: NCT00920309
Title: Rapamycin as Treatment for ADPKD: The Role of Biomarkers in Predicting a Response to Therapy
Brief Title: Rapamycin as Treatment for Autosomal Dominant Polycystic Kidney Disease (ADPKD): The Role of Biomarkers in Predicting a Response to Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study was stopped after larger studies published in the NEJM failed to show a benefit in treating ADPKD
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC#0903004934
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal Dominant Polycystic Kidney Disease; rapamycin; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapamycin (Experimental): Drug: Rapamycin
  Other Names:
  sirolimus The starting dose of rapamycin will be 1 mg daily. The dose will be increased as needed to achieve a 24 hour trough level of 4-6 ng/ml.
  Interventions: Drug: Rapamycin
- Standard of Care-Placebo (Placebo Comparator): Standard of Care
  Interventions: Other: Standard of Care-Placebo

INTERVENTIONS:
Drug: Rapamycin — The starting dose of rapamycin will be 1 mg daily. The dose will be increased as needed to achieve a 24 hour trough level of 4-6 ng/ml.
  Other Names: sirolimus
  Arms: Rapamycin
Other: Standard of Care-Placebo
  Arms: Standard of Care-Placebo

SUMMARY:
Currently the only approved use for rapamycin (sirolimus) is for immunosuppression after renal transplantation.

This trial is designed to determine whether rapamycin is safe and effective treatment for patients with polycystic kidney disease (ADPKD). Patients will be followed by volumetric magnetic resonance imaging (MRI) to observe for change in kidney (and cyst) size. Blood and urine samples will also be collected to evaluate for change in biomarkers with treatment.

DETAILED DESCRIPTION:
This is a 2 year, open label trial to evaluate the role of rapamycin as treatment for ADPKD. Patients will be randomized 2:1 to the rapamycin arm or to standard therapy. The dose of rapamycin will be adjusted so that patients obtain 24 trough levels of 4-6ng/ml. There will be a volumetric MRI measurement at the start and end of the treatment period. Patients will be monitored every 4 months throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* adult ADPKD patients aged 18-70
* combined kidney volume >1200 ml
* estimated creatinine clearance >60 ml/min
* absence of implanted ferromagnetic objects

Exclusion Criteria:

* Age >70
* uncontrolled hyperlipidemia
* Proteinuria >500 mg/day
* unstable cerebral aneurysm
* active coronary artery disease
* diagnosis of another systemic condition affecting kidney function (ie: diabetes, hepatitis B or C, HIV)
* diagnosis of cancer other than skin cancer
* pregnancy or lactation
* presence of implanted ferromagnetic objects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neera K Dahl, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapamycin | Standard of Care-Placebo
Started | 14 | 7
Completed | 14 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapamycin | Standard of Care-Placebo | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 20
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Kidney Volume (mL)
Time Frame: 2 years
Population: Outcome Measures were not analyzed due to study termination
Groups:
- Rapamycin: The study was terminated before any enrolled patients were treated for 2 years.
Arm/Group | Rapamycin | Standard of Care-Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Glomerular Filtration Rate (Kidney Function)
Time Frame: 2 years
Population: Outcome measures were not analyzed due to study termination
Arm/Group | Rapamycin | Standard of Care-Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study occurred over a 1 year time period which was on adverse events were collected. This study was terminated early.
Arm/Group | Rapamycin | Standard of Care-Placebo
Serious Adverse Events (participants affected / at risk) | 3/14 | 0/7
Other Adverse Events (participants affected / at risk) | 14/14 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rapamycin (N=14) | Standard of Care-Placebo (N=7)
Hyperglycemia (Endocrine disorders) | 1 | 0
Flank Pain (General disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rapamycin (N=14) | Standard of Care-Placebo (N=7)
Cellulitis of the ear (Infections and infestations) | 1 | 0
Upper Respiratory Infesion (Infections and infestations) | 1 | 0
Heart Palipitations with Hypertension (Cardiac disorders) | 1 | 0
Edema/Weight gain (Vascular disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Apothous Ulcer (Infections and infestations) | 2 | 0
Increased Liver Function Test (Hepatobiliary disorders) | 2 | 0
Hyperglycemia (Endocrine disorders) | 1 | 0
Emesis/Diarrhea (Gastrointestinal disorders) | 2 | 0
Impaired Depth Perception (Nervous system disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (General disorders) | 1 | 0
Sinus Headache (General disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Abscess (Skin and subcutaneous tissue disorders) | 2 | 0
Allergic Rhinitis (General disorders) | 1 | 0
Dysuria (Endocrine disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Epistaxis (General disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Left Hip Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pedal Edema (Vascular disorders) | 1 | 0
Hives (Skin and subcutaneous tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ear/Neck Pain (General disorders) | 1 | 0
Bloating/Flatulence (Gastrointestinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Facial Sensitivity (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No